CLINICAL TRIAL: NCT01080508
Title: Analysis of the Spirometry Pattern in Esophageal Intubation
Brief Title: Spirometry in Esophageal Intubation
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: Lazarus 001
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Intubation
Keywords: pressure pattern; esophageal and tracheal ventilation.; esophageal intubation.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group 1: asa 1&2 patients
  Interventions: Other: tracheal ventilation with regular tube
- group 2: asa 1&2 patients
  Interventions: Other: ventilation after intubation with special tube

INTERVENTIONS:
Other: tracheal ventilation with regular tube — Description of the pressure waveforms during tracheal ventilation
  Groups: group 1
Other: ventilation after intubation with special tube — Description of the pressure waveforms during esophageal ventilation
  Groups: group 2

SUMMARY:
The primary objective of the study is to describe the pressure patterns during esophageal and tracheal ventilation and to validate the diagnostic algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients, requiring total anesthesia for a surgical procedure where the use of the easytube could be indicated.

Exclusion Criteria:

* ASA III
* Expected difficulty for oral intubation.
* Expected operation time >3 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I & II patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Determination of the sensitivity and specificity of the algorithm to detect esophageal intubation. | during intubation

SECONDARY OUTCOMES:
Pressure pattern of ventilation in esophageal and tracheal ventilation. | during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Alain F kalmar, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, University of Groningen, the Netherlands, Groningen, Netherlands

REFERENCES:
- [Derived] Kalmar AF, Absalom A, Monsieurs KG. A novel method to detect accidental oesophageal intubation based on ventilation pressure waveforms. Resuscitation. 2012 Feb;83(2):177-82. doi: 10.1016/j.resuscitation.2011.10.009. Epub 2011 Oct 30. PMID 22044726